CLINICAL TRIAL: NCT02029131
Title: Effects of a Home-based Exercise Program on Low Back Pain in Employees
Brief Title: Exercise and Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Responsible Party: Principal Investigator, Sven Haufe, Dr. rer. medic., Hannover Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SpoMed Low Back
Record Dates: First submitted 2014-01-03; First posted 2014-01-07 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Healthy Volunteers With and Without Chronic Low Back Pain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Controls (No Intervention)

INTERVENTIONS:
Behavioral: Exercise — Educated exercise training for the trunk 3 times per week, each for 20 min. Recommendation of additional fitness courses as offered by the local healthy insurance company.
  Arms: Exercise

SUMMARY:
Evaluation of the effectiveness of an individually educated exercise program for the lower back at home in employees over a period of 20 weeks.

We hypothesize that regular exercise for the lower back results in greater improvements of low back strengths compared to controls.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* age between 18 and 67 years

Exclusion Criteria:

* beeing currently involved in an exercise program for the lower back
* known drug or alcohol abuse
* any disease that excludes the participation in an exercise program
* clinical relevant acute or chronic infections
* pregnant women

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Back strength (kg) | At baseline and after 20 weeks
  Assessed with the back-check 607 (Dr. WOLFF Sports and Prevention)

SECONDARY OUTCOMES:
Strenght at lateral flexion of the trunk (kg) | At baseline and after 20 weeks
  Assessed with the back-check 607 (Dr. WOLFF Sports and Prevention)
Oswestry Low Back Pain Disability Score | At baseline and after 20 weeks
  Assessed with the Oswestry Low Back Pain Disability questionaire
Pain (scale) | At baseline and after 20 weeks
  Assessed with the visual analog scale
Quality of life (score) | At baseline and after 20 weeks
  Assessed with the short form 36 questionaire
Work ability index (score) | At baseline and afetr 20 weeks
  Assessed with the WAI questionaire
Physical activity (score) | At baseline and after 20 weeks
  Assessed with the "Freiburger activity questionaire"
Fat mass and fat-free mass (kg) | At baseline and after 20 weeks
  Assessed with Bio Impedance Analysis
sick days (numbers) | At baseline and after 20 weeks
  sick days at work will be assessed for the 20 weeks of the active intervention and the whole year the intervention is conducted

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Bayerle P, Kerling A, Kuck M, Rolff S, Boeck HT, Sundermeier T, Ensslen R, Tegtbur U, Lauenstein D, Bothig D, Bara C, Hanke A, Terkamp C, Haverich A, Stiesch M, de Zwaan M, Haufe S, Nachbar L. Effectiveness of wearable devices as a support strategy for maintaining physical activity after a structured exercise intervention for employees with metabolic syndrome: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2022 Feb 10;14(1):24. doi: 10.1186/s13102-022-00409-1. PMID 35144658